CLINICAL TRIAL: NCT00248352
Title: GLUCOSE : Glucose Lowering by Usual Care Or Specialized Endocrinology Team
Brief Title: A Study Comparing Standard Care for Diabetes to Case-Managed Care for Diabetes in Patients With Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Sanofi (Industry); Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: Glucose 101
Record Dates: First submitted 2005-11-01; First posted 2005-11-03 (Estimated); Last update posted 2007-10-26 (Estimated); Status verified 2007-10

CONDITIONS: Diabetes Mellitus, Type 2; Coronary Disease
Keywords: Coronary Artery Disease; Diabetes Mellitus; Type 2; Chronic Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Disease; Coronary Artery Disease; Diabetes Mellitus; Chronic Disease | interventions — Referral and Consultation; Endocrinologists

INTERVENTIONS:
Behavioral: Consultation with Endocrinologist
Behavioral: Counseling from Dietician
Behavioral: Counseling from Diabetes Educator

SUMMARY:
The purpose of this study is to compare two ways to treat patients with Type 2 Diabetes, Standard Care or Case-Managed Care.

In-Patient Standard Care is guided by the assigned cardiologist and Out-Patient Standard Care by the existing diabetes care givers.

Case-Managed care involves a consult with an endocrinologist and counseling from a diabetic educator and a dietician.

DETAILED DESCRIPTION:
Patients with diabetes have a higher incidence of coronary artery disease and a worsened cardiac prognosis. Death from cardiovascular disease accounts for about 70% of all diabetes-related deaths (Booth, 2003). Diabetes is also a common problem among hospitalized cardiac patients. In Ontario, from 1995 to 1997, nearly 1/3 of the 104,471 patients admitted for acute myocardial infarction had diabetes (Booth, 2003). In these patients, hyperglycemia remains a marker for poor outcome despite improvements in coronary care (Wahab, 2002; Capes, 2000).

Several important questions regarding the diabetes care of cardiac patients admitted to hospital wards are yet to be answered. First, it is not known if better glycemic control during the ward phase of hospitalization in itself improves short-term outcomes. Second, assuming that short-term glycemic control is beneficial, it is not known which interventions are effective in accomplishing this. Third, assuming that putting more resources into the management and education of patients with diabetes will translate into long term benefits, it is not known whether this should be done during the "window of opportunity" provided by a cardiac admission or whether this intervention will be more effective if it is deferred until after discharge.

These critical treatment dilemmas have prompted the proposal for the GLUCOSE Pilot Study, a randomized, controlled study to examine the effectiveness of case-managed diabetes care using a multidisciplinary team approach in patients with diabetes admitted to manage concomitant ischemic heart disease. We have designed this protocol to study the effectiveness of case-managed diabetes care by a specialized endocrinology team and compare it to usual care as delivered by the attending cardiologist. Patients will be randomized to specialized endocrinology care or usual care at the time of their admission to the ward. The short-term outcome will be glycemic control of cardiac patients with diabetes while they are admitted to a cardiology ward. In order to compare this with a more typical model of post-discharge care, patients will be re-randomized at the time of discharge into case-managed or usual care groups. The long-term (primary) outcome will be glycemic control and risk factor reduction at 6 months. This factorial design will allow us to compare several treatment models and determine which is the most efficient and effective way to achieve the best long-term diabetes control and risk factor management in our patients.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus, type 2, as defined by at least one of the following:

  * Previous diagnosis of diabetes
  * two glucose levels consistent with diabetes (fasting glucose >7.0 mmol/L or random glucose >11.0 mmol/L )
  * HbA1C > 6.5% using DCCT standardized methods And

Coronary Disease, as defined by at least one of the following:

* Admitting diagnosis of acute coronary syndrome defined by 2/3 of typical history, enzyme changes, dynamic ECG changes
* Prior history of acute coronary syndrome defined as above
* Previously documented myocardial infarction
* Previous coronary revascularization procedure
* Coronary artery disease defined by coronary angiography
* Exercise or persantine nuclear perfusion imaging positive for ischemia

Exclusion Criteria:

* Refusal to enter the study
* Inability to understand consent forms and provide informed consent
* Anticipated length of non-ICU hospital stay less than 48 hours
* Diabetes Mellitus, type 1

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2005-02; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Change in HbA1C at 6 months post discharge compared to baseline measure obtained at the time of discharge
Change in 10 year cardiac risk as estimated by the UKPDS risk engine at 6 months post discharge compared to baseline measures obtained at time of discharge

SECONDARY OUTCOMES:
Percentage of patients with capillary blood glucose values within a target range of > 4.0 mmol/L to < 10.0 mmol/L during hospitalization
Number of patients with one or more episodes of hypoglycemia defined as capillary blood glucose measurements < 4.0 mmol/L
Number of patients with one or more episodes of persistent hyperglycemia defined as three consecutive capillary blood glucose measurements > 15.0 mmol/L
Number of patients on prognosis improving medications (ACE inhibitor, ARB, Lipid Lowering Agents)
Number of patients having death, MI, stroke, recurrent ischemic event or readmission to hospital
Length of stay
Risk factor control at 6 months post discharge:
Blood pressure control, defined as percentage of patients within 2003 Canadian Diabetes Association Clinical Practice Guidelines (December 2003)
Lipid levels within 2003 Canadian Diabetes Association Clinical Practice Guidelines (December 2003)
Percentage of patients, who were smokers at time of index admission, who have quit
Exercise history
Patient satisfaction with inpatient diabetes management as measured by a standardized questionnaire administered prior to discharge
Diabetes self-care as assessed by questionnaire
Quality of life as assessed by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Richard F. Davies, M.D., Principal Investigator — University of Ottawa Heart Instittue; Janine Malcolm, M.D., Principal Investigator — Ottawa Hospital
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Bhattacharyya A, Christodoulides C, Kaushal K, New JP, Young RJ. In-patient management of diabetes mellitus and patient satisfaction. Diabet Med. 2002 May;19(5):412-6. doi: 10.1046/j.1464-5491.2002.00716.x. PMID 12027930
- [Background] Booth G, Fang J. Acute complications of Diabetes: In Hux JE, Booth GL, Slaughter PM, Laupacis A (eds.). Diabetes in Ontario: An ICES Practice Atlas. Institute for Clinical Evaluative Sciences. 2003:2.21-2.51.
- [Background] Brown SA. Meta-analysis of diabetes patient education research: variations in intervention effects across studies. Res Nurs Health. 1992 Dec;15(6):409-19. doi: 10.1002/nur.4770150603. PMID 1448572
- [Background] Canadian Diabetes Association Clinical Practice Guidelines Expert Committee; Cheng AY. Canadian Diabetes Association 2013 clinical practice guidelines for the prevention and management of diabetes in Canada. Introduction. Can J Diabetes. 2013 Apr;37 Suppl 1:S1-3. doi: 10.1016/j.jcjd.2013.01.009. Epub 2013 Mar 26. No abstract available. PMID 24070926
- [Background] Capes SE, Hunt D, Malmberg K, Gerstein HC. Stress hyperglycaemia and increased risk of death after myocardial infarction in patients with and without diabetes: a systematic overview. Lancet. 2000 Mar 4;355(9206):773-8. doi: 10.1016/S0140-6736(99)08415-9. PMID 10711923
- [Background] Cavan DA, Hamilton P, Everett J, Kerr D. Reducing hospital inpatient length of stay for patients with diabetes. Diabet Med. 2001 Feb;18(2):162-4. doi: 10.1046/j.1464-5491.2001.00420.x. PMID 11251683
- [Background] Clement S. Diabetes self-management education. Diabetes Care. 1995 Aug;18(8):1204-14. doi: 10.2337/diacare.18.8.1204. No abstract available. PMID 7587866
- [Background] Davies M, Dixon S, Currie CJ, Davis RE, Peters JR. Evaluation of a hospital diabetes specialist nursing service: a randomized controlled trial. Diabet Med. 2001 Apr;18(4):301-7. doi: 10.1046/j.1464-5491.2001.00470.x. PMID 11437861
- [Background] Egan BM, Greene EL, Goodfriend TL. Nonesterified fatty acids in blood pressure control and cardiovascular complications. Curr Hypertens Rep. 2001 Apr;3(2):107-16. doi: 10.1007/s11906-001-0021-y. PMID 11276390
- [Background] Furnary AP, Zerr KJ, Grunkemeier GL, Starr A. Continuous intravenous insulin infusion reduces the incidence of deep sternal wound infection in diabetic patients after cardiac surgical procedures. Ann Thorac Surg. 1999 Feb;67(2):352-60; discussion 360-2. doi: 10.1016/s0003-4975(99)00014-4. PMID 10197653
- [Background] Gaede P, Vedel P, Larsen N, Jensen GV, Parving HH, Pedersen O. Multifactorial intervention and cardiovascular disease in patients with type 2 diabetes. N Engl J Med. 2003 Jan 30;348(5):383-93. doi: 10.1056/NEJMoa021778. PMID 12556541
- [Background] Golden SH, Peart-Vigilance C, Kao WH, Brancati FL. Perioperative glycemic control and the risk of infectious complications in a cohort of adults with diabetes. Diabetes Care. 1999 Sep;22(9):1408-14. doi: 10.2337/diacare.22.9.1408. PMID 10480501
- [Background] Hux JE, Tang M. Patterns of prevalence and incidence of diabetes: In Hux JE, Booth GL, Slaughter APM, Laupacis (eds). Diabetes in Ontario: An ICES Practice Atlas. Institute for Clinical and Evaluative Sciences. 2003:1.1-1.18.
- [Background] Janes JM, Bradley C, Rees A. Preferences for, and improvements in aspects of quality of life (QoL) with, insulin lispro in a multiple injection regimen. Diabetologia. 1997;40, Suppl. 1:A353.
- [Background] Renders CM, Valk GD, Griffin SJ, Wagner EH, Eijk Van JT, Assendelft WJ. Interventions to improve the management of diabetes in primary care, outpatient, and community settings: a systematic review. Diabetes Care. 2001 Oct;24(10):1821-33. doi: 10.2337/diacare.24.10.1821. PMID 11574449
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] van den Berghe G, Wouters P, Weekers F, Verwaest C, Bruyninckx F, Schetz M, Vlasselaers D, Ferdinande P, Lauwers P, Bouillon R. Intensive insulin therapy in critically ill patients. N Engl J Med. 2001 Nov 8;345(19):1359-67. doi: 10.1056/NEJMoa011300. PMID 11794168
- [Background] Wahab NN, Cowden EA, Pearce NJ, Gardner MJ, Merry H, Cox JL; ICONS Investigators. Is blood glucose an independent predictor of mortality in acute myocardial infarction in the thrombolytic era? J Am Coll Cardiol. 2002 Nov 20;40(10):1748-54. doi: 10.1016/s0735-1097(02)02483-x. PMID 12446057
- [Background] Lawlor D, Vandewater D, Ur E. Diabetes. Case management. Can Nurse. 2002 Jan;98(1):27-30. No abstract available. PMID 11845552
- [Background] Levetan CS, Passaro MD, Jablonski KA, Ratner RE. Effect of physician specialty on outcomes in diabetic ketoacidosis. Diabetes Care. 1999 Nov;22(11):1790-5. doi: 10.2337/diacare.22.11.1790. PMID 10546009
- [Background] Levetan CS, Salas JR, Wilets IF, Zumoff B. Impact of endocrine and diabetes team consultation on hospital length of stay for patients with diabetes. Am J Med. 1995 Jul;99(1):22-8. doi: 10.1016/s0002-9343(99)80100-4. PMID 7598138
- [Background] Malmberg K. Prospective randomised study of intensive insulin treatment on long term survival after acute myocardial infarction in patients with diabetes mellitus. DIGAMI (Diabetes Mellitus, Insulin Glucose Infusion in Acute Myocardial Infarction) Study Group. BMJ. 1997 May 24;314(7093):1512-5. doi: 10.1136/bmj.314.7093.1512. PMID 9169397
- [Background] Malmberg K, Ryden L, Efendic S, Herlitz J, Nicol P, Waldenstrom A, Wedel H, Welin L. Randomized trial of insulin-glucose infusion followed by subcutaneous insulin treatment in diabetic patients with acute myocardial infarction (DIGAMI study): effects on mortality at 1 year. J Am Coll Cardiol. 1995 Jul;26(1):57-65. doi: 10.1016/0735-1097(95)00126-k. PMID 7797776
- [Background] Queale WS, Seidler AJ, Brancati FL. Glycemic control and sliding scale insulin use in medical inpatients with diabetes mellitus. Arch Intern Med. 1997 Mar 10;157(5):545-52. PMID 9066459
- [Background] Polonsky WH, Earles J, Smith S, Pease DJ, Macmillan M, Christensen R, Taylor T, Dickert J, Jackson RA. Integrating medical management with diabetes self-management training: a randomized control trial of the Diabetes Outpatient Intensive Treatment program. Diabetes Care. 2003 Nov;26(11):3048-53. doi: 10.2337/diacare.26.11.3048. PMID 14578238
- [Background] Manzella D, Carbonella M, Ragno E, Passariello N, Grella R, Paolisso G. Relationship between autonomic cardiac activity, beta-cell function, anthropometrics and metabolic indices in type II diabetics. Clin Endocrinol (Oxf). 2002 Aug;57(2):259-64. doi: 10.1046/j.1365-2265.2002.01596.x. PMID 12153606
- [Background] Koproski J, Pretto Z, Poretsky L. Effects of an intervention by a diabetes team in hospitalized patients with diabetes. Diabetes Care. 1997 Oct;20(10):1553-5. doi: 10.2337/diacare.20.10.1553. PMID 9314634